CLINICAL TRIAL: NCT01976286
Title: A Pilot Study Comparing the Efficacy of Glycolic Acid Peels vs. Salicylic Acid Peels for the Treatment of Melasma: A Randomized Control Trial
Brief Title: A Pilot Study Testing Salicylic Acid Peels Versus Glycolic Acid Peels for the Treatment of Melasma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU84250
Record Dates: First submitted 2013-10-15; First posted 2013-11-05 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Melanosis
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Salicylic Acid Peels (Active Comparator): Salicylic Acid and Glycolic Acid Chemical Peels are skin treatments used to correct uneven texture and color by removing dead cells from the skin's top layer.
  Interventions: Other: Salicylic Acid Peels
- Glycolic Acid Peels (Active Comparator): Salicylic Acid and Glycolic Acid Chemical Peels are skin treatments used to correct uneven texture and color by removing dead cells from the skin's top layer.
  Interventions: Other: Glycolic Acid Peels

INTERVENTIONS:
Other: Salicylic Acid Peels
  Arms: Salicylic Acid Peels
Other: Glycolic Acid Peels
  Arms: Glycolic Acid Peels

SUMMARY:
The purpose of this study is to find out the safety and effectiveness of Glycolic Acid Chemical Peels compared to Salicylic Acid Chemical Peels for the treatment of melasma.

DETAILED DESCRIPTION:
Participants in this study will be patients who are clinically diagnosed with at least a 2 x 2 cm patch of melasma on each side of their face (forehead or cheek). One half of the subject's face will be randomly selected to receive 4 treatments of 30% glycolic acid peels and the other half of the face will receive 4 treatments of 30% salicylic acid peels/ weeks 0, 4, 8, and 12. Follow up visit will be at week 16. This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years or older
2. Subjects with at least a 2 x 2 cm patch of melasma on each side of the face (forehead or cheek)
3. Subjects in general good health
4. Subjects must be willing and able to understand and provide informed consent for the use of their tissue and communicate with the investigator
5. Subjects must be willing to not apply other treatment options for melasma during the course of the study

Exclusion Criteria:

1. Subjects under 18 years of age
2. Subjects who are pregnant and/or lactating
3. Subjects who are unable to understand the protocol or to give informed consent
4. Subjects diagnosed with mental illness
5. Subjects who have concurrent active uncontrolled disease to facial area (i.e uncontrolled acne)
6. Subjects who have had a chemical peel in the past 3 months
7. Subjects who have used a prescribed retinoid in the past 3 months
8. Subjects with a bleeding disorder
9. Subjects with a history of abnormal wound healing
10. Subjects with a history of abnormal scarring

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in best overall cosmetic appearance (right side or left side better)rated by a blinded dermatologist from baseline to week 16 | 1 hour at baseline and week 16
  The primary outcome was a blinded rating of the treatment area (Salicylic Acid Peels Versus Glycolic Acid Peels) with the best overall cosmetic appearance. A dermatologist will blindly evaluate the treated areas of each side from live subjects at baseline and on the final follow up visit (week 16).

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States